CLINICAL TRIAL: NCT06390670
Title: The Effect of Colostrum Bovinum Supplementation on Upper Respiratory Tract Infections Rate and Selected Immunological Biomarkers in Trained Athletes: a Randomized, Crossover, Placebo-controlled, Double-blind Trial
Brief Title: The Effect of Colostrum Bovinum Supplementation in Endurance Athletes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Nutricia Foundation (Other); Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Prof Dr hab., PhD, Poznan University of Physical Education
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDS2022_0002
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Sports Nutrition; Biochemical Markers; Exercise Performance; Aerobic Capacity; Supplementation
Keywords: Sports dietetics; Immunomodulation; Immunodepression; Physical capacity; Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COL supplementation (Experimental): The experimental procedure for each participant in this group includes a 12-week period of COL supplementation.
  The entire study protocol included familiarization and 4 main visits to the laboratory (T1-T4; pre/post supplementation with COL and PLA). After the familiarization, enrolled volunteers were randomly assigned (stratified randomization) to the treatment order by an impartial biostatistician. A 4-week washout period was introduced between treatments. The main study protocol included body mass and composition evaluation, 3 saliva and blood samplings (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) and 2 exercise protocols during each of T1-T4 study visit (interspaced with 50 min of passive rest and 10 min of warm-up before the second exercise test). All testings were performed in the morning hours at the same time for the participant, to avoid physiological diurnal fluctuations in measured saliva and blood outcomes.
  Interventions: Dietary Supplement: Colostrum Bovinum supplementation
- PLA treatment (Placebo Comparator): The experimental procedure for each participant in this group includes a 12-week period of PLA supplementation.
  The entire study protocol included familiarization and 4 main visits to the laboratory (T1-T4; pre/post supplementation with COL and PLA). After the familiarization, enrolled volunteers were randomly assigned (stratified randomization) to the treatment order by an impartial biostatistician. A 4-week washout period was introduced between treatments. The main study protocol included body mass and composition evaluation, 3 saliva and blood samplings (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) and 2 exercise protocols during each of T1-T4 study visit (interspaced with 50 min of passive rest and 10 min of warm-up before the second exercise test). All testings were performed in the morning hours at the same time for the participant, to avoid physiological diurnal fluctuations in measured saliva and blood outcomes.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Colostrum Bovinum supplementation — In the experimental procedure each athlete was supplemented with a chronic dose of 25 g/day of COL. Supplement was particularly prepared for the study from a first post-delivery milking and had a high content of IgG (60%; certified Colostrum Bovinum; Agrapak, Poland). The COL was provided in the powder form and were taken twice a day (12.5 g in the morning and 12.5 g in the afternoon). Participants were instructed to dissolved each portion of the COL supplement in 250 mL of plain water.
  Arms: COL supplementation
Other: Placebo treatment — In the control procedure each athlete was supplemented with a chronic dose of 25 g/day of placebo (PLA). PLA was particularly prepared for the study, and was an isoenergetic/isomacronutrient product (high quality protein) prepared for the trial (Agrapak, Poland). The PLA was provided in the powder form and were taken twice a day (12.5 g in the morning and 12.5 g in the afternoon). Participants were instructed to dissolved each portion of the PLA preparation in 250 mL of plain water.
  Arms: PLA treatment

SUMMARY:
The purpose of this study was to verify the effect of chronic 12-week high-dose Colostrum Bovinum (COL) and placebo (PLA) supplementation on immunological, hematological and biochemical markers, as well as physical capacity and discipline-specific exercise performance in endurance athletes, in a randomized, double-blind, placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Colostrum Bovinum (COL) is a substance produced naturally by mammary glands of mammals for 24-72 h after calving. The significant impact of COL supply on the development of the immune system of the calves has led to the beginning of the use of COL supplementation in humans to improve their immune functions. Intense physical activity suppresses immunity up to several hours after training, which is known as the "open window". Due to large volumes of intense efforts that athletes of endurance sports disciplines undergo (especially swimmers and triathletes), they are at high risk for immunological disorders, especially upper respiratory tract infections (URTI), such as the common cold. There are limited studies applying to the supplementation of COL in athletes in order to positively affect immune system. Currently, there is only one systematic review and meta-analysis of 5 randomized controlled trials showing that oral supplementation of COL can reduce the incidence rate of URTI days and episodes in athletes. In terms of immunological biomarkers, there are conflicting studies. In one of them, a 33% increase in salivary secretory (SIgA) was observed after 2-week of 20g COL supplementation. In the other study, the use of a 12-week period of supplementation of a chocolate drink containing 12 g COL in a group of runners led to a 79% increase in resting SIgA. On the contrary, some of the studies found no significant difference in SIgA between COL-supplemented and placebo groups. However, latter studies found beneficial effects of COL intake on the stimulation of neutrophil oxidative burst, blunting the prolonged exercise-induced decrease in in vivo immune responsiveness to a novel antigen and the reduction in exercise-induced muscle damage and markers of inflammation.

Based on these results, it can be concluded that COL supplementation may have a beneficial effect on the immune system of athletes. However, it is required to conduct well-controlled standardized studies, which can be characterized by the sufficient dose and period of the effective supplementation, to identify markers of immune system adequate for evaluation of the response in case of such stimulation. Therefore, the study aimed to examine the effect of chronic 12-week high-dose COL and placebo (PLA) supplementation on immunological, hematological and biochemical markers, as well as physical capacity and discipline-specific exercise performance in endurance athletes, in a randomized, double-blind, placebo-controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* a good health condition without chronic health disorders,
* a valid and up-to-date medical certificate confirming the athlete's ability to practice sports,
* at least 5 years of triathlon/swimming training experience,
* regular participation in triathlon/swimming competitions on at least national level.

Exclusion Criteria:

* allergy to cow's milk proteins,
* lactose intolerance,
* any autoimmune diseases,
* reporting symptoms of infection or taking any medication (longer than 3 days) for 4 weeks before the enrollment to the study protocol.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in saliva secretory IgA (SIgA) concentration after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the saliva SIgA concentration (μg/mL) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in upper respiratory tract infections rate during COL supplementation and PLA treatment. | 12 weeks during COL supplementation and PLA treatment.
  Assessment of the upper respiratory tract infections (URTI) rate by measuring rate ratio of URTI days, rate ratio of episodes of URTI and duration of URTI episodes during assigned interventions (during COL and PLA treatment).

SECONDARY OUTCOMES:
Changes in white blood cells count after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the white blood cells (neutrophils, monocytes, lymphocytes, granulocytes, neutrophils:lymphocytes ratio) (count/L) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in white blood cells differential after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the white blood cells (neutrophils, monocytes, lymphocytes, granulocytes) (%) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in blood Tumour Necrosis Factor alpha (TNF- α), Interleukin-6 (IL-6), and Interleukin-10 (IL-10) cytokines after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the TNF- α, IL-6, and IL-10 cytokines concentration (pg/mL) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in blood Interferon-gamma cytokine (IFN-γ) after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the IFN-γ concentration (ng/L) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in blood immunoglobulins A (IgA), M (IgM), G (IgG) after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the IgA, IgM, IgG immunoglobulins concentration (g/L) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in blood immunoglobulins D (IgD) and E (IgE) after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the IgD, IgE immunoglobulins concentration (IU/mL) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in salivary bacterial load after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the salivary bacterial load (count/mL) at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in blood natural killer cells after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the natural killer cells (count) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in aerobic capacity and incremental rowing test (IRT) performance measured by maximum workload at exhaustion after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the aerobic capacity and IRT performance (measured by maximum workload at exhaustion in Watts) was carried out by an incremental rowing test to exhaustion at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in aerobic capacity measured by maximal oxygen uptake after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the aerobic capacity (maximal oxygen uptake in mL/min/kg) was carried out by an incremental rowing test to exhaustion at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in the discipline-specific exercise performance after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the exercise performance (time trial performance in min) was carried out during a swimming-specific performance test consisting of eight 100-meter-long sections to swim through, of which the sections I-III were performed at level of 75% maximal effort [ME, determined during the familiarization visit], IV-V at 85% ME, VI at 90% ME, VII at 95% ME and VIII at 100% ME), with 1 to 2.5 min of recovery between sections. The test was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in lactate concentration (mmol/L) before and after exercise tests after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the lactate concentration (mmol/L) was performed at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA) from fingertip capillary blood: a) before and 3-min after the IRT to exhaustion; b) during recovery break between sections of the discipline-specific exercise performance test and 3-min after the last section at four main visits to the laboratory; and c) 1 h after the cessation of the second exercise protocol (the discipline-specific exercise performance test).
Changes in heart rate during exercise protocols. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the heart rate (bpm) during both exercise protocols was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in blood C-C motif chemokines Ligand 2 (CCL2), 3 (CCL3), 4 (CCL4), and C-X-C motif chemokine ligand 9 (CXCL9) after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the CCL2, CCL3, CCL4, CXCL9 chemokines concentration (pg/mL) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in nutritional status indices (concentration of total protein and albumin, glucose) (g/dL) after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the nutritional status indices (concentration of total protein, albumin, glucose) concentration (g/dL) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Changes in Insulin-like Growth Factor 1 (IGF-1) (ng/mL) after COL supplementation and PLA treatment. | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of the IGF-1 concentration (ng/mL) in blood at three time-points (resting [REST]; 3 min [POST-EX] and 60 min after completion of the second test exercise [REC]) was carried out at four main visits to the laboratory (T1-T4; before/after supplementation with COL and PLA).
Analysis of body composition (fat-free mass, fat mass). | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of body composition (fat-free mass, fat mass) (kg) was carried out before the execution of exercise protocols on each research visit.
Analysis of body composition (% fat-free mass, % fat mass). | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of body composition (% of fat-free mass, and % of fat mass) was carried out before the execution of exercise protocols on each research visit.
Analysis of body composition (total body water). | Before and after 12 weeks of COL suplementation and PLA treatment.
  Assessment of body composition (total body water) (%) was carried out before the execution of exercise protocols on each research visit.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, Prof., PhD, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Department of Sports Dietetics, Poznan University of Physical Education, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Durkalec-Michalski K, Glowka N, Podgorski T, Wochna K, Wozniewicz M, Nowaczyk PM. Twelve-Week Colostrum Bovinum Supplementation Supports Aerobic Capacity but has No Effect on Body Composition in Endurance-Trained Males: A Randomized Placebo-Controlled Crossover Study. Eur J Sport Sci. 2025 May;25(5):e12288. doi: 10.1002/ejsc.12288. PMID 40254930